CLINICAL TRIAL: NCT00364416
Title: ADHERE (Acute Decompensated Heart Failure National Registry) Longitudinal Module-Registry of Advanced Heart Failure Patients at High Risk for Rehospitalization
Brief Title: Longitudinal Registry for Advanced Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Scios, Inc. (Industry)
Responsible Party: Sr. Director, Clinical Team Leader, Scios
Other Study IDs: CR005212
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Heart Failure, Congestive; Heart Decompensation
Keywords: Heart Failure, congestive; Heart decompensation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001
  Interventions: Other: Any treatment used to treat CHF

INTERVENTIONS:
Other: Any treatment used to treat CHF — Clinical Outcomes of Chronic Decompensated Heart Failure patients

SUMMARY:
The purpose of this study is to gather information to better understand the characteristics, medical management techniques and outcomes of patients with chronic severe Heart Failure (HF).

DETAILED DESCRIPTION:
This objectives of this observational registry are: to assess changes in patient quality of life as a function of medical management and disease progression as measured by the rate of death and rehospitalization, and assist with the optimization of heart failure (HF) management by providing information on the use of therapies proven to be effective and to describe practices of standard of care for chronic treatment of symptoms of HF outside the hospital and during hospitalization for acute episode with intravenous vasoactive medication (drugs which affect the blood vessels and muscle of the heart). Additional information which will be gathered include patient characteristics (age, sex, race, medical history, symptoms), infusion setting, type of medication, dose and frequency of medication and worsening of congestive heart failure disease. Participants in the study receive an unique patient-specific identifier and all available data will be analyzed. Observational Study - No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Age older than or equal to 18 years at the time of entry into the Registry
* Severe symptoms of HF at rest with marked limitation of physical activity continuously for at least 60 days prior to inclusion in the Registry
* Patient has been hospitalized 2 times in the past 12 months with a primary diagnosis of HF
* Patient's HF is refractory or relatively refractory to usual non-IV medications, as defined by having received one of the two following regimens for the treatment of HF in that last 60 days: 2 complete IV infusions, each lasting at least 2 hours, of either vasoactive (drugs having an effect on veins or arteries) or inotrope medications (drugs that makes the heart works better), or 3 IV diuretic (drugs that increase the elimination of urine) treatments

Exclusion Criteria:

* History of any organ transplantation
* Patient is expected to die within the next 5 days
* Patient is seen for consultation or evaluation only, and is unlikely to receive follow-up care at the participating clinic/hospital
* Participation in a clinical study of the drug Natrecor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HF who present with severe symptoms limiting their physical activities at rest
Sampling Method: Non-Probability Sample
Enrollment: 1466 (Actual)
Dates: Start 2002-10; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome are length of hospitalization and/or time to death | Patients data are collected for 2 years. Data are collected for all scheduled and unscheduled office visits, and each hospitalization. Individual patient questionnaires are completed at baseline and every 3 months thereafter.

SECONDARY OUTCOMES:
Evaluation of medication and other treatment received | every 3 months
Evaluation of laboratory results | evey 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.